CLINICAL TRIAL: NCT07028801
Title: A Randomized, Blinded, Parallel Controlled, Non-inferiority Design Phase III Clinical Trial to Evaluate the Immunogenicity and Safety of Freeze-dried Human Rabies Vaccine (Human Diploid Cells) Administered to Participants Aged 10 to 60 Years With Different Immunization Schedules
Brief Title: Clinical Trial of Freeze-dried Human Rabies Vaccine (Human Diploid Cells)
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ningbo Rongan Biological Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: AIM2301-Ⅲ-01
Record Dates: First submitted 2025-06-03; First posted 2025-06-19 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Rabies
MeSH Terms: conditions — Rabies

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- group 1 (Experimental): The Participants received 1 dose of Rabies Vaccine（Human Diploid Cell）for Human Use,Freeze-dried each at day 0, 3, 7, 14 and 28, with a total of 5 doses.
  Interventions: Biological: Freeze-dried human rabies vaccine (human diploid cells)
- group 2 (Experimental): The Participants received 1 dose of Rabies Vaccine（Human Diploid Cell）for Human Use,Freeze-dried each at day 0, 3, 7, and14, with a total of 4 doses.
  Interventions: Biological: Freeze-dried human rabies vaccine (human diploid cells)
- group 3 (Experimental): The Participants received 1 dose of Rabies Vaccine（Human Diploid Cell）for Human Use,Freeze-dried each at day 0, 3, 7 and 28, with a total of 4 doses.
  Interventions: Biological: Freeze-dried human rabies vaccine (human diploid cells)
- group 4 (Experimental): The Participants received 2 doses of Rabies Vaccine（Human Diploid Cell）for Human Use,Freeze-dried on day 0, 1 dose on day 7 and 1 dose on day 21, a total of 4 doses.
  Interventions: Biological: Freeze-dried human rabies vaccine (human diploid cells)
- group 5 (Active Comparator): The Participants received 1 dose of Rabies Vaccine（Human Diploid Cell）for Human Use,Freeze-dried each at day 0, 3, 7, 14 and 28, with a total of 5 doses.
  Interventions: Biological: Freeze-dried human rabies vaccine (human diploid cells)

INTERVENTIONS:
Biological: Freeze-dried human rabies vaccine (human diploid cells) — This vaccine is produced by Ningbo Rongyu Biopharmaceutical Co., LTD. Participants will be administered 5 doses of freeze-dried human rabies vaccine (human diploid cells) by intramuscular injection.
  Receive 1 dose on day 0, 3, 7, 14 and 28, total 5 doses
  Arms: group 1
Biological: Freeze-dried human rabies vaccine (human diploid cells) — This vaccine is produced by Ningbo Rongyu Biopharmaceutical Co., LTD. Participants will be administered 4 doses of freeze-dried human rabies vaccine (human diploid cells) by intramuscular injection.
  Receive 1 dose on day 0, 3, 7 and 14, total 4 doses
  Arms: group 2
Biological: Freeze-dried human rabies vaccine (human diploid cells) — This vaccine is produced by Ningbo Rongyu Biopharmaceutical Co., LTD. Participants will be administered 4 doses of freeze-dried human rabies vaccine (human diploid cells) by intramuscular injection.
  Receive 1 dose on day 0, 3, 7 and 28, total 4 doses
  Arms: group 3
Biological: Freeze-dried human rabies vaccine (human diploid cells) — This vaccine is produced by Ningbo Rongyu Biopharmaceutical Co., LTD. Participants will be administered 4 doses of freeze-dried human rabies vaccine (human diploid cells) by intramuscular injection.
  Receive 2 dose on day 0, 1 dose on day 7 and 21, total 4 doses
  Arms: group 4
Biological: Freeze-dried human rabies vaccine (human diploid cells) — This vaccine is produced by Chengdu Kanghua Biological Products Co., LTD Participants will be administered 5 doses of freeze-dried human rabies vaccine (human diploid cells) by intramuscular injection
  Receive 1 dose on day 0, 3, 7, 14and 28, total 5 doses
  Arms: group 5

SUMMARY:
The Phase 3 clinical trial of freeze-dried human rabies vaccine (human diploid cells) adopted a randomized, blinded, parallel control,non-inferiority design,and administered vaccines to participants aged 10 to 60 years with different immunization schedules (5-dose schedule group, two simple 4-dose schedule groups, and 2-1-1 schedule group) to evaluate the immunogenicity and safety of the vaccine.

DETAILED DESCRIPTION:
The trial will use a randomized, blinded, parallel-group, non-inferiority design. A total of 3000 participants will be planned to be randomly assigned in a 1:1:1:1:1 ratio to the 5-dose control vaccine schedule, the 5-dose experimental vaccine schedule, the simple 4-dose experimental vaccine schedule 1, the simple 4-dose experimental vaccine schedule 2, and the 2-1-1 trial vaccine schedule, with 600 participants in each group, including 100 participants aged 10 to 17 years and 500 participants who will be 18-60 years old. Immunogenicity visits will be scheduled for all participants: (1) 5-dose schedule group: before dose 1, day 7 (before dose 3), day 14 (7 after dose 3, before dose 4), day 28 (14 after dose 4, before dose 5), day 42 (14 days after the full schedule); (2) Simple four-dose schedule group 1: before dose 1, day 14 (7 days after dose 3 and before dose 4), day 28 (14 days after the full dose), and day 42 (28 days after the full schedule); (3) Simple four-dose schedule group 2: before dose 1, day 14 (7 days after the third dose), day 28 (before the fourth dose), and day 42 (14 days after the full schedule); (4) 2-1-1 schedule group: before dose 1, day 7 (before the third dose), day 14 (7 days after the third dose) and day 35 (14 days after the full schedule). If the vaccination is delayed, the blood collection time will be postponed according to the vaccination time of the corresponding dose.

A total of 1200 participants in the immune persistence subgroup (including 200 participants aged 10-17 years and 1000 participants aged 18-60 years) will be selected. Blood samples will be collected at 3 months and 6 months after the full schedule of vaccination to evaluate the immune persistence. The first 40% of participants in the 10 to 17 years of age group and the 18 to 60 years of age group enrolled at each site will be selected as participants in the immune persistence subgroup.

All participants will be observed for safety events that will occur from the first dose through 30 days after the full schedule and for SAEs and pregnancy events that will be reported from the first dose through 6 months after the full schedule.

ELIGIBILITY:
Inclusion Criteria:

* (1) The participants' ages range from 10 to 60 years old (≥10 years old and <61 years old).

  (2) Participants aged 10 to 17 and their guardians can provide valid identification documents, and participants aged 18 to 60 can provide their own valid identification documents.

  (3) Participants aged 10 to 17 and their guardians, as well as participants aged 18 to 60, can sign the informed consent form voluntarily to participate in the trial, fully understand the trial procedures, the risks of participating in the trial, and other intervention measures that can be chosen if they do not participate in the trial, etc.

  (4) Possess basic reading and writing skills, and be capable of reading, understanding and filling in diary cards and contact cards; (5) Female participants with fertility must also meet the following conditions: 1) They have taken effective contraceptive measures within two weeks prior to participating in this trial; 2) Have no plans to have children within 6 months from the start of participating in this trial until the full vaccination. 3) Understand and agree to take effective contraceptive measures during the trial period (from the first dose to within 6 months after the full vaccination). Effective contraceptive measures include: condoms (for men), intrauterine devices, oral contraceptives (excluding emergency contraceptives), sterilization, abstention, injection or implantable contraception, sustained-release local contraceptives, hormone patches, diaphragms, cervical caps, etc. External ejaculation and safe period contraception are not regarded as effective contraceptive measures.

Exclusion Criteria:

* For the standards marked with *, if the participants have the circumstances stipulated in the standard, the visit can be rescheduled when they no longer have these circumstances

  1. After inquiry, it is found that there is a history of rabies vaccination or the use of passive immunization preparations for rabies virus.
  2. There was a history of injury from rabies virus-susceptible animals (such as cats and dogs) before the first dose of vaccination;
  3. The axillary body temperature of the participants on the day of enrollment was ≥37.3℃*;
  4. Women who have a positive urine pregnancy trial before vaccination (on the day of vaccination), or who, after assessment, cannot rule out the possibility of pregnancy or are breastfeeding;
  5. Hypertension that cannot be controlled by medication, such as systolic blood pressure ≥160mmHg and/or diastolic blood pressure ≥100mmHg for participants aged 18 years and above before enrollment;
  6. Allergy to any component of the vaccine used in the trial, such as human albumin, sucrose, or maltose;
  7. Those with a history of severe allergies in the past, such as anaphylactic shock, allergic laryngeal edema, allergic purpura, local allergic necrosis reaction (Arthus reaction), severe urticaria, allergic bronchitis, acquired angioedema, etc.
  8. Has been diagnosed with congenital or acquired immune system diseases, such as the Human Immunodeficiency Virus. HIV infection, lymphoma, leukemia, systemic lupus erythematosus, rheumatoid arthritis, juvenile rheumatoid arthritis, inflammatory bowel disease or other immune diseases that the researcher deems likely to affect the trial assessment;
  9. Known or suspected of having serious diseases, including severe respiratory diseases, liver and kidney diseases, cardiovascular and cerebrovascular diseases, malignant tumors, and other chronic diseases that are poorly controlled, etc.
  10. Abnormal coagulation function (such as deficiency of coagulation factors, coagulation disorders, abnormal platelets) or coagulation disorders diagnosed by a doctor;
  11. Anplenia or functional anplenia, as well as anplenia or splenectomy caused by any circumstances;
  12. Previous or current clearly diagnosed neurological or mental disorders (including but not limited to dementia, schizophrenia, bipolar disorder, etc.) or confirmed epilepsy, convulsions, as well as other neurological or mental disorders that the researcher deems unsuitable for participation in this trial;
  13. It is planned to receive such treatment from the first dose of vaccination to 30 days after the full vaccination course, such as long-term systemic glucocorticoid therapy (used continuously for 2 weeks or more, at a dose of ³2mg/kg/ day or ³20mg/ day prednisone or equivalent doses); Local medications (such as ointments, eye drops, inhalants or nasal sprays) are allowed;
  14. Have received or plan to receive immunoenhancers or inhibitors, immunoglobulins or blood-related products throughout the trial period within 3 months prior to enrollment;
  15. Have received attenuated live vaccines within 14 days before enrollment, and subunit vaccines or inactivated vaccines within 7 days *;
  16. Within 3 days before enrollment, have suffered from acute diseases or be in the acute attack stage of chronic diseases *;
  17. Antipyretic, analgesic and antihistamine drugs were used within 3 days before enrollment.
  18. Currently participating in or planning to participate in other clinical trials during this clinical trial;
  19. According to the researcher's judgment, due to various medical, psychological, social conditions or other circumstances contrary to the trial protocol, or the participants' inability to comply with the requirements of the trial protocol.

Ages: 10 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 3000 (Estimated)
Dates: Start 2025-07-31 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Antibody SCR for the 5-dose schedule group of the trial vaccine and the 5-dose schedule group of the control vaccine | 14 days after the first dose
  Antibody seroconversion rates in the 5-dose schedule group of the trial vaccine and the 5-dose control vaccine group.
Antibody GMC for the 5-dose schedule group of the trial vaccine and the 5-dose schedule group of the control vaccine | 14 days after the first dose
  Antibody Geometric Mean Concentration in the 5-dose schedule group of the trial vaccine and the 5-dose control vaccine group.
Antibody SCR for the simple 4-dose schedule group 1 of the trial vaccine and the 5-dose schedule group of the control vaccine | 14 days after the first dose
  Antibody seroconversion rates in the simple 4-dose schedule group 1 of the trial vaccine and in the 5-dose group of the control vaccine.
Antibody GMC for the simple 4-dose schedule group 1 of the trial vaccine and the 5-dose schedule of the control vaccine | 14 days after the first dose
  Antibody Geometric Mean Concentration in the simple 4-dose schedule group 1 of the trial vaccine and in the 5-dose group of the control vaccine.
Antibody SCR for the simple 4-dose schedule group 2 of the trial vaccine and the 5-dose schedule group of the control vaccine | 14 days after the first dose
  Antibody seroconversion rates in the simple 4-dose schedule group 2 of the trial vaccine and in the 5-dose group of the control vaccine.
Antibody GMC for the simple 4-dose schedule group 2 of the trial vaccine and the 5-dose schedule group of the control vaccine | 14 days after the first dose
  Antibody Geometric Mean Concentration in the simple 4-dose schedule group 2 of the trial vaccine and in the 5-dose group of the control vaccine.
Antibody SCR for the 2-1-1 schedule group of the trial vaccine and the 5-dose schedule group of the control vaccine | 14 days after the first dose
  Antibody seroconversion rates in the 2-1-1 schedule group of the trial vaccine and in the 5-dose group of the control vaccine.
Antibody GMC for the 2-1-1 schedule group of the trial vaccine and the 5-dose schedule group of the control vaccine | 14 days after the first dose
  Antibody Geometric Mean Concentration in the 2-1-1 schedule group of the trial vaccine and in the 5-dose group of the control vaccine.
Antibody SCR for the 5-dose schedule group of the trial vaccine and the 5-dose schedule group of the control vaccine | 14 days after full vaccination
  Antibody seroconversion rates in the 5-dose schedule group of the trial vaccine and the 5-dose control vaccine group.
Antibody SCR for the simple 4-dose schedule group 1 of the trial vaccine and the 5-dose schedule group of the control vaccine | 14 days after full vaccination
  Antibody seroconversion rates in the simple 4-dose schedule group 1 of the trial vaccine and in the 5-dose group of the control vaccine.
Antibody SCR for the simple 4-dose schedule group 2 of the trial vaccine and the 5-dose schedule group of the control vaccine | 14 days after full vaccination
  Antibody seroconversion rates in the simple 4-dose schedule group 2 of the trial vaccine and in the 5-dose group of the control vaccine.
Antibody SCR for the 2-1-1 schedule group of the trial vaccine and the 5-dose schedule group of the control vaccine | 14 days after full vaccination
  Antibody seroconversion rates in the 2-1-1 schedule group of the trial vaccine and in the 5-dose group of the control vaccine.

CONTACTS AND LOCATIONS:
Locations (1):
- Henan Provincial Center for Disease Control and Prevention, Zhengzhou, Henan, China